CLINICAL TRIAL: NCT07281677
Title: Immunogenicity and Safety of Sequential Bivalent and 9-Valent Human Papillomavirus Vaccine Immunization in Girls Aged 9-14 Years
Brief Title: Immunogenicity and Safety of Sequential 2vHPV-9vHPV Vaccination in Girls Aged 9-14 Years
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Shenyu Wang, Deputy Director, Department of Immunization Program, Zhejiang Provincial Center for Disease Control and Prevention
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2025-065-01
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: HPV Infection
Keywords: HPV; bivalent HPV vaccine; 9-valent HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Participants will receive one dose of the bivalent HPV vaccine, followed by two doses of the 9-valent HPV vaccine six months later[2v-9v-9v (0, 6m, 12m)].
  Interventions: Biological: bivalent HPV vaccine; Biological: 9-valent HPV vaccine
- Group B (Experimental): Participants will receive one dose of the 9-valent HPV vaccine sequentially 6 months after receiving one dose of the bivalent HPV vaccine[2v-9v(0, 6m)].
  Interventions: Biological: bivalent HPV vaccine; Biological: 9-valent HPV vaccine
- Control (Active Comparator): Participants will receive two doses of the 9-valent HPV vaccine directly[9v-9v(0, 6m)].
  Interventions: Biological: 9-valent HPV vaccine
- External control (Other): Participants will receive two doses of the bivalent HPV vaccine directly[2v-2v(0, 6m)].
  Interventions: Biological: bivalent HPV vaccine

INTERVENTIONS:
Biological: bivalent HPV vaccine — Bivalent HPV vaccine produced by Shanghai Zerun Biotechnology Co.,Ltd. or Wantai BioPharm.
  Arms: External control; Group A; Group B
Biological: 9-valent HPV vaccine — 9-valent HPV vaccine is produced by Wantai BioPharm or Merck Sharp & Dohme LLC.
  Arms: Control; Group A; Group B

SUMMARY:
This study aims to assess the immunogenicity and safety of a sequential 2vhpv to 9vhpv immunization schedule in girls aged 9-14 years

DETAILED DESCRIPTION:
A post-marketing study is being conducted in Zhejiang Province to evaluate the immunogenicity and safety of a sequential 2vhpv to 9vhpv immunization schedule in girls aged 9-14 years. The study plans to recruit 300 healthy participants, who will be randomly assigned in a 1:1:1 ratio to three groups. In Experimental Group A, participants will receive one dose of the bivalent HPV vaccine followed six months later by two doses of the 9-valent HPV vaccine. In Experimental Group B, participants will receive one dose of the 9-valent HPV vaccine six months after a single dose of the bivalent HPV vaccine. The control group will receive two doses of the 9-valent HPV vaccine at a six-month interval. Venous blood samples will be collected before the first dose, one month before and after each dose of the 9-valent vaccine, and at 12 and 24 months after full immunization to assess HPV vaccine-type-specific neutralizing antibodies.

In addition, 100 healthy girls will be enrolled as an external control group receiving two doses of the bivalent vaccine, with blood samples collected before each dose and at 1, 12, and 24 months post-vaccination to assess HPV vaccine-type-specific neutralizing antibodies.

ELIGIBILITY:
Inclusion Criteria

* Have not received any HPV vaccine products.
* Girls aged 9 to 14 years.
* Reside permanently at the research site. Both the participant and her legal guardian have voluntarily agreed to participate, have signed the informed consent form, understand and agree to comply with the study protocol, and are able to complete all scheduled blood collections and follow-up visits.

Exclusion Criteria

* Suspected or confirmed fever (≥38.5°C) within 72 hours prior to enrollment, or axillary temperature >37.0°C on the day of enrollment.
* HIV infection or other immunocompromising conditions.
* Presence of acute illness or being in the acute phase of a chronic disease.
* History of severe allergic reactions to any component of the study vaccine or to previous vaccinations.
* Contraindications to intramuscular injection, such as thrombocytopenia, coagulation disorders, or current anticoagulant therapy.
* Receipt of non-live vaccines within 14 days or live attenuated vaccines within 28 days prior to HPV vaccination in this study.
* Receipt of blood or blood-derived products within 3 months prior to enrollment, or planned use within 6 months from the first vaccination to completion of the full vaccination schedule.
* Any disease or condition deemed by the investigator to place the participant at unacceptable risk, prevent adherence to study requirements, or interfere with the assessment of vaccine responses.

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-12-20 (Estimated); Study Completion 2029-11-13 (Estimated)

PRIMARY OUTCOMES:
Seropositive rate of the vaccination | Before the first vaccine, before and 1 month after each dose of the 9-valent vaccine, and 12 and 24 months after the entire vaccination course. External Control Group: Before each vaccine, and 1, 12, and 24 months after the entire vaccination course
  The percentage of participants with positive antibody against vaccine-specific HPV
Seroconversion rate of the vaccination | Before the first vaccine, before and 1 month after each dose of the 9-valent vaccine, and 12 and 24 months after the entire vaccination course. External Control Group: Before each vaccine, and 1, 12, and 24 months after the entire vaccination course
  The proportion of participants who are determined to have seroconversion of Vaccine-specific HPV antibody
Geometric mean concentration (GMC) | Before the first vaccine, before and 1 month after each dose of the 9-valent vaccine, and 12 and 24 months after the entire vaccination course. External Control Group: Before each vaccine, and 1, 12, and 24 months after the entire vaccination course
  The GMC of vaccine-specific HPV antibody
Geometric mean increase (GMI) | Before the first vaccine, before and 1 month after each dose of the 9-valent vaccine, and 12 and 24 months after the entire vaccination course. External Control Group: Before each vaccine, and 1, 12, and 24 months after the entire vaccination course
  The GMI of vaccine-specific HPV antibody

SECONDARY OUTCOMES:
Description of AE; Incidence of AR and SAE | within 30 minutes and within 30 days after vaccination (AE/AR); within 6 months after the entire vaccination course
  Describe AE according to study group, site of occurrence, severity, and relevance; calculate the incidence rates of AR and SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Shenyu Wang, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Jinyun center for Disease Control and Prevention, Lishui, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No